CLINICAL TRIAL: NCT04805892
Title: Open Label, Single-Center Study Utilizing BIOZEK COVID-19 Antigen Rapid Test as Compared to Standard Testing Technique. Test Performed by a Professional Versus Self-collection and Standard of Care
Brief Title: Study Utilizing BIOZEK COVID-19 Antigen Rapid Test.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mach-E B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: #Biozek-ARTC-US
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Diagnostic Test: BIOZEK COVID-19 Antigen Rapid Test — The BIOZEK COVID-19 Antigen Rapid Test is used for the detection of SARS-CoV-2 antigens in nasopharyngeal swab specimens from individuals who are suspected of having COVID-19.

SUMMARY:
This is a research study to evaluate the Sensitivity and Specificity of BIOZEK COVID-19 Antigen Rapid Test on samples collected by a healthcare professional versus self-collection; and to perform analysis to compare results. In addition, to obtain RT-PCR test results, performed prior to enrollment, and compare all three results.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be ≥18 years of age and have had an RT-PCR test performed prior to enrollment.

Subjects must be able to understand and willingly sign a written informed consent. Additionally, participants need to meet at least 1 of the criteria listed below:

* Currently experiencing symptoms of COVID-19.
* Be clinically diagnosed or suspected to have COVID-19.
* Recent past (3 weeks) exhibited symptoms of COVID-19.
* Be capable of performing a self-collection of a nasopharyngeal sample with use of nasal swab kit.
* Interacted with a COVID-19 positive individual.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria may not be enrolled in this study:

* Cannot perform self-collection of a nasopharyngeal sample with use of nasal swab kit.
* Have a deviated nasal septum.
* Cognitively impaired individuals resulting in the inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mobile Covid Services LLC, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site study was performed by Mobile Covid Services, a COVID-19 testing concierge service. Enrollment and testing took place at the subject's home. The Enrollment population consisted of symptomatic and asymptomatic subjects scheduled for an appointment to perform an RT-PCR test for SARS-CoV-2 as the standard of care procedure.
Groups:
- BIOZEK COVID-19 Antigen Rapid Test: BIOZEK COVID-19 Antigen Rapid Test as compared to standard testing technique. Test performed by a professional versus self-collection and standard of care.
Period: Overall Study
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test
Number analyzed (Participants) | 84
Age, Customized [Count of Participants; unit: Participants]
  Age 18 - 85 years | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 13
  More than one race | 39
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 84

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of BIOZEK COVID-19 Antigen Rapid Test on a Sample Collected by Healthcare Professionals.
Description: The Biozek Antigen Rapid Tests performed by the trained study personnel on the samples collected by the trained study personnel. Sensitivity was calculated using (TP/TP+FN)*100% formula.
  Specificity was calculated using (TN/TN+FP)*100% formula.
Time Frame: 1 visit, up to 2 hours
Population: One subject was excluded from the analysis due to inconclusive results.
Measure: Number; unit: percentage - Sensitivity and specificity
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test
Number analyzed (Participants) | 83
percentage - Sensitivity and specificity
  Sensitivity - Test performed by trained study personnel: number analyzed (Participants) | 33
  Sensitivity - Test performed by trained study personnel | 100
  Specifity - Test performed by trained study personnel: number analyzed (Participants) | 50
  Specifity - Test performed by trained study personnel | 98

2. Secondary Outcome: Sensitivity and Specificity of BIOZEK COVID-19 Antigen Rapid Test on Self - Collected Samples.
Description: The Biozek Antigen Rapid Tests self-performed performed by the subject on the self - collected samples by the subjects. Sensitivity was calculated using (TP/TP+FN)*100% formula.
  Specificity was calculated using (TN/TN+FP)*100% formula.
Time Frame: 1 visit, up to 2 hours
Population: One subject was excluded from the analysis due to inconclusive results.
Measure: Number; unit: percentage - Sensitivity and specificity
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test
Number analyzed (Participants) | 83
percentage - Sensitivity and specificity
  Sensitivity - Test performed by the subject | 100
  Specificity - Test performed by the subject | 98

ADVERSE EVENTS:
Time Frame: 1 visit - up to 2 hours
Groups:
- Biozek Covid-19 Antigen Test: No adverse events were reported.
Arm/Group | Biozek Covid-19 Antigen Test
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT04805892/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT04805892/ICF_001.pdf